CLINICAL TRIAL: NCT03273751
Title: The Effect of Remote Ischemic Preconditioning on Kidney Function in Patients Undergoing Partial Nephrectomy : A Randomized Controlled Trial
Brief Title: The Effect of Remote Ischemic Preconditioning on Kidney Function in Patients Undergoing Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1707-087-870
Record Dates: First submitted 2017-09-03; First posted 2017-09-06 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Renal Neoplasm; Renal Injury
Keywords: Remote Ischemic Preconditioning; Partial nephrectomy; Acute kidney injury
MeSH Terms: conditions — Kidney Neoplasms; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, parallel group, controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators and outcome assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Preconditioning (RIPC) (Experimental): Four cycles of upper arm ischemia/reperfusion
  Interventions: Procedure: Remote Ischemic Preconditioning
- Sham control (Sham Comparator): Placement of a blood pressure cuff around upper arm without inflation.
  Interventions: Procedure: Sham control

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — After induction of anesthesia, RIPC consisted of four 5-min cycles of limb ischemia induced by a blood pressure cuff placed on the upper arm and inflated to 250 mmHg, with an intervening 5 min of reperfusion during which the cuff was deflated.
  Other Names: RIPC
  Arms: Remote Ischemic Preconditioning (RIPC)
Procedure: Sham control — After induction of anesthesia, sham control consisted of the placement of a blood pressure cuff on the upper arm with no inflation during the surgery.
  Arms: Sham control

SUMMARY:
This study is intended to evaluate the renal protective effect of Remote Ischemic Preconditioning (RIPC) in patients undergoing partial nephrectomy. Half of the enrolled subjects will receive 4 cycles of brief ischemia on the upper arm after anesthesia induction and prior to the surgery, while the other half will not receive this treatment as a control group.

DETAILED DESCRIPTION:
Remote Ischemic Preconditioning (RIPC) is the concept of mitigating ischemia-reperfusion injury to target organs by a brief episode of ischemia-reperfusion of the limb. The protective effect of RIPC on major organs has been demonstrated in an animal study, but its clinical efficacy has not yet been established.

The kidney is a typical organ vulnerable to ischemic injury, and the renal protective effect of RIPC can be expected. There have been many reports of renal protective effects of RIPC in cardiac and vascular surgery. On the other hand, few studies have investigated the effect of RIPC during partial nephrectomy in which ischemia-reperfusion injury can occur during the surgery.

In this study, the investigators will evaluate the effect of RIPC in patients undergoing partial nephrectomy to prevent renal impairment and improve the prognosis after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled to undergo open, laparoscopic, or robot-assisted laparoscopic partial nephrectomy
* Normal contralateral renal function was defined as split renal function of >40% as determined by preoperative Tc-99m DiethyleneTriamine Pentaacetic Acid (DTPA) kidney scan
* Written informed consent

Exclusion Criteria:

* Peripheral vascular disease involving upper extremities or lower extremities
* Severe cardiopulmonary diseases (valvular or ischemic heart disease, heart failure, chronic obstructive pulmonary disease)
* Hepatic failure, renal failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Serum creatinine level | Postoperative day 1
  Postoperative serum creatinine levels as an index of kidney damage

SECONDARY OUTCOMES:
The incidence of acute kidney injury (AKI) | Within 7 days after surgery
  The incidence of AKI according to the serum creatinine diagnostic criteria of Kidney Disease Improving Global outcomes (KDIGO) Clinical Practice Guideline for AKI
Serum creatinine level | 1 hour after surgery
  Postoperative serum creatinine levels as an index of kidney damage
Serum creatinine level | Postoperative day 3
  Postoperative serum creatinine levels as an index of kidney damage
Serum creatinine level | 2 weeks after surgery
  Postoperative serum creatinine levels as an index of kidney damage
estimated glomerular filtration rate (eGFR) | 1 hour after surgery
  eGFR is obtained by the formula of Isotope Dilution Mass Spectrometry (IDMS) Modification of Diet in Renal Disease (MDRD).
estimated glomerular filtration rate (eGFR) | Postoperative day 1
  eGFR is obtained by the formula of Isotope Dilution Mass Spectrometry (IDMS) Modification of Diet in Renal Disease (MDRD).
estimated glomerular filtration rate (eGFR) | Postoperative day 3
  eGFR is obtained by the formula of Isotope Dilution Mass Spectrometry (IDMS) Modification of Diet in Renal Disease (MDRD).
estimated glomerular filtration rate (eGFR) | 2 weeks after surgery
  eGFR is obtained by the formula of Isotope Dilution Mass Spectrometry (IDMS) Modification of Diet in Renal Disease (MDRD).
Regional oxygen saturation (rSO2) of the contralateral kidney of the operated side | 5 min after the induction of anesthesia (baseline)
  Renal rSO2 of the contralateral kidney of the operated side is monitored with Near-infrared spectroscopy.
Regional oxygen saturation (rSO2) of the contralateral kidney of the operated side | 30 minutes after induction of anesthesia
  Renal rSO2 of the contralateral kidney of the operated side is monitored with Near-infrared spectroscopy.
Regional oxygen saturation (rSO2) of the contralateral kidney of the operated side | 60 minutes after induction of anesthesia
  Renal rSO2 of the contralateral kidney of the operated side is monitored with Near-infrared spectroscopy.
Regional oxygen saturation (rSO2) of the contralateral kidney of the operated side | 90 minutes after induction of anesthesia
  Renal rSO2 of the contralateral kidney of the operated side is monitored with Near-infrared spectroscopy.
Urine creatinine level | Postoperative day 1
  Urine creatinine level
Urine creatinine level | 2 weeks after surgery
  Urine creatinine level
Urine microalbumin | Postoperative day 1
  Urine microalbumin
Urine microalbumin | 2 weeks after surgery
  Urine microalbumin
Urine beta-2 microglobulin | Postoperative day 1
  Urine beta-2 microglobulin
Urine beta-2 microglobulin | 2 weeks after surgery
  Urine beta-2 microglobulin
Urine N-acetyl-beta-D-glucosaminidase | Postoperative day 1
  Urine N-acetyl-beta-D-glucosaminidase
Urine N-acetyl-beta-D-glucosaminidase | 2 weeks after surgery
  Urine N-acetyl-beta-D-glucosaminidase
Glomerular filtration rate measured by scintigraphy | preoperative baseline
  Glomerular filtration rate measured by technetium diethylene triamine pentacetic acid (99mTc-DTPA) radionuclide scintigraphy
Glomerular filtration rate measured by scintigraphy | 6 months after surgery
  Glomerular filtration rate measured by technetium diethylene triamine pentacetic acid (99mTc-DTPA) radionuclide scintigraphy
Glomerular filtration rate measured by scintigraphy | 12 months after surgery
  Glomerular filtration rate measured by technetium diethylene triamine pentacetic acid (99mTc-DTPA) radionuclide scintigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang J, Chen Y, Dong B, Kong W, Zhang J, Xue W, Liu D, Huang Y. Effect of remote ischaemic preconditioning on renal protection in patients undergoing laparoscopic partial nephrectomy: a 'blinded' randomised controlled trial. BJU Int. 2013 Jul;112(1):74-80. doi: 10.1111/bju.12004. Epub 2013 Mar 4. PMID 23452148
- [Background] Zarbock A, Schmidt C, Van Aken H, Wempe C, Martens S, Zahn PK, Wolf B, Goebel U, Schwer CI, Rosenberger P, Haeberle H, Gorlich D, Kellum JA, Meersch M; RenalRIPC Investigators. Effect of remote ischemic preconditioning on kidney injury among high-risk patients undergoing cardiac surgery: a randomized clinical trial. JAMA. 2015 Jun 2;313(21):2133-41. doi: 10.1001/jama.2015.4189. PMID 26024502
- [Background] Zhang L, Diao Y, Chen G, Tanaka A, Eastwood GM, Bellomo R. Remote ischemic conditioning for kidney protection: A meta-analysis. J Crit Care. 2016 Jun;33:224-32. doi: 10.1016/j.jcrc.2016.01.026. Epub 2016 Feb 10. PMID 26936039
- [Derived] Hur M, Park SK, Shin J, Choi JY, Yoo S, Kim WH, Kim JT. The effect of remote ischemic preconditioning on serum creatinine in patients undergoing partial nephrectomy: a study protocol for a randomized controlled trial. Trials. 2018 Sep 4;19(1):473. doi: 10.1186/s13063-018-2820-3. PMID 30180887